CLINICAL TRIAL: NCT02497222
Title: Pilot Study of RNS60 in Allergen-induced Bronchconstriction
Brief Title: Pilot Study of RNS60 in Allergen-induced Bronchoconstriction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 01.1.1.H4
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — RNS60; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RNS60 (Experimental): RNS60 4 ml, inhaled twice daily by nebulization for 21 days.
  Interventions: Drug: RNS60
- Normal Saline (Placebo Comparator): Normal Saline 4 ml, inhaled twice daily by nebulization for 21 days.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: RNS60
  Arms: RNS60
Drug: Normal Saline
  Arms: Normal Saline

SUMMARY:
This study evaluates the use of RNS60 in the treatment of asthma examining regional improvements in inflammation using PET imaging. All subjects will be treated with both RNS60 and placebo in a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with mild asthma (as defined by the National Institutes of Health 2002 Guidelines for the Diagnosis and Management of Asthma (2)) with symptoms more than 2 times a week but less than once per day with normal FEV1 (> 80% predicted).
* Clinical history of allergic symptoms to cat or dust mite allergen and demonstrated skin reactivity.
* Subjects must have a lifetime total of less than 5 pack years with no smoking in the previous 5 years.
* Willing and able to give informed consent and adhere to the study protocol requirements.
* Expressed the desire to participate in the study in an interview with the principal investigator (PI).
* Age between 18 and 50 years.

Exclusion Criteria:

* Women of childbearing potential who are documented to be pregnant (based on blood beta-human chorionic gonadotropin [HCG] testing) or who are nursing.
* The presence of spontaneous asthmatic episode or clinical evidence of upper respiratory tract infection within the previous 6 weeks.
* Participation in research study involving a drug or biologic during the 30 days prior to the study.
* Intolerance to albuterol, atropine, or lidocaine.
* Antihistamines within 7 days of the screening visit.
* Known exposure to agents that are associated with pulmonary disease (i.e. asbestos, silica).
* Presence of other known pulmonary disease, coronary disease, congestive heart failure, ventricular arrhythmias, history of a cerebrovascular accident, renal failure (or creatinine > 1.5, if known), history of anaphylaxis, cirrhosis, diabetes mellitus or presence of a significant disease, which in the opinion of the PI would pose a significant risk for the subject or confound the results of the study.
* Use of systemic steroids, increased use of inhaled steroids, use of beta blockers and monoamine oxidase (MAO) inhibitors or a visit for an asthma exacerbation within 1 month of the screening visit.
* A history of asthma-related respiratory failure requiring intubation.
* A history of hospitalization for asthma.
* Subjects with a high possibility of poor compliance with the study as judged by the PI.
* Unresponsive to bronchodilator agents.
* Quantitative skin prick test at or below a dilution level of standardized cat allergen extract of 1:2048 (4.88 BAU/ml) for subjects being challenged with cat allergen.
* Quantitative skin prick test at or below a dilution level of standardized mite allergen extract of 1:2048 (4.88 AU/ml) for subjects being challenged with either mite allergen.
* Subjects who, by participating in any research study, will have a cumulative radiation dose exceeding 50 mSv in the previous year.
* Contraindication to Methacholine challenge testing (heart attack or stroke in last 3 months, uncontrolled hypertension, or known aortic aneurysm).
* Body Mass Index (BMI) > 32.
* Individuals with known allergy or hypersensitivity to FDG will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
18F-FDG uptake rate | 21 days
  Comparison of fluorodeoxyglucose (18F-FDG) uptake rate in subjects before and after inhalation of RNS60 or placebo

SECONDARY OUTCOMES:
Regional VA and Vdef volume | 21 days
  Comparison of regional ventilation (VA) and ventilation defective areas (Vdef) volume in subjects before and after inhalation of RNS60 or placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States